CLINICAL TRIAL: NCT05020678
Title: A Phase 1 Study of NKX019, a CD19 Chimeric Antigen Receptor Natural Killer (CAR NK) Cell Therapy, in Subjects With B-cell Malignancies
Brief Title: NKX019, Intravenous Allogeneic Chimeric Antigen Receptor Natural Killer Cells (CAR NK), in Adults With B-cell Cancers
Status: Active, not recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: Nkarta, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: NKX019-101
Record Dates: First submitted 2021-08-20; First posted 2021-08-25 (Actual); Last update posted 2024-12-24 (Actual); Status verified 2024-12

CONDITIONS: Lymphoma, Non-Hodgkin; B-cell Acute Lymphoblastic Leukemia; Large B-cell Lymphoma; Mantle Cell Lymphoma; Indolent Lymphoma; Waldenstrom Macroglobulinemia; Chronic Lymphocytic Leukemia; Small Lymphocytic Lymphoma; Aggressive Lymphoma; Large-cell Lymphoma
Keywords: CD19; CAR; Allogeneic; Natural killer; ACR; NKX019; IL15; Interleukin 15; NK cell; Cell Therapy; Immunotherapy; Adoptive cell therapy; r/r NHL; r/r B-ALL; r/r MCL; r/r IL; r/r WM; r/r CLL; r/r SLL; Aggressive lymphoma; Indolent lymphoma; LCL
MeSH Terms: conditions — Lymphoma, Non-Hodgkin; Burkitt Lymphoma; Lymphoma, Mantle-Cell; Waldenstrom Macroglobulinemia; Leukemia, Lymphocytic, Chronic, B-Cell; Dendritic Cell Sarcoma, Interdigitating

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- NKX019 - CAR NK cell therapy (Experimental): All subjects will receive fludarabine/cyclophosphamide lymphodepletion followed by 3 weekly doses of NKX019 on Day 0, 7, and 14 of a 28-day cycle. Combination cohorts (if opened) will additionally receive rituximab with each cycle.
  Interventions: Biological: NKX019

INTERVENTIONS:
Biological: NKX019 — NKX019 is an investigational allogeneic CAR NK product targeting CD19 on cells. The starting dose of NKX019 in Part 1 is 3 × 10^8 NK cells (6 × 10^6/kg for patients < 50 kg) administered as 3 weekly doses. Part 2 (dose expansion cohorts) will use the maximum tolerated dose (MTD) or recommended Phase 2 dose (RP2D) of NKX019 as determined in Part 1.

SUMMARY:
This is a single arm, open-label, multi-center, Phase 1 study to determine the safety and tolerability of an experimental therapy called NKX019 (allogeneic CAR NK cells targeting CD19) in patients with relapsed/refractory non-Hodgkin lymphoma (NHL), chronic lymphocytic leukemia (CLL) or B cell acute lymphoblastic leukemia (B-ALL)

DETAILED DESCRIPTION:
This is a dose-finding study of NKX019 and will be conducted in 2 parts:

Part 1: dose finding utilizing a "3+3" enrollment schema and safety lead-in to confirm dose for NKX019 in combination with rituximab expansion cohorts (as applicable) Part 2: dose expansion to further evaluate safety and tolerability, cellular kinetics, pharmacodynamics and anti-tumor response in expansion cohorts of patients with large B cell lymphoma (LBCL), mantle cell lymphoma (MCL), indolent lymphoma (IL), Waldenström macroglobulinemia (WM), CLL/ small lymphocytic lymphoma (SLL), and B-ALL.

ELIGIBILITY:
Inclusion Criteria:

General:

Eastern Cooperative Oncology Group (ECOG) performance status ≤1

• Disease Related:

* Have a histologically or cytologically confirmed diagnosis of r/r B cell NHL or CLL or B-ALL as defined by WHO 2016 classification
* Subjects who received prior CD19/CD20-directed therapy must have disease that remains CD19+ and/or CD20+ respectively
* Have measurable disease
* Have received ≥2 lines of therapy except subjects with MCL, CAR T Naïve cohorts and WM, who must have received at least 1 prior line of therapy
* Have received a combination of an anti CD20 monoclonal antibody and cytotoxic chemotherapy for subjects with NHL
* Received:

  * BTKi for subjects with MCL, CLL/SLL, WM, and other indications where a BTKi is approved
  * Venetoclax for subjects with CLL/SLL
  * Tyrosine kinase inhibitor for subjects with Philadelphia chromosome (Ph+) B-ALL
* Not responded or relapsed within 12 months of completion of their prior line of therapy, with the exception of a newly diagnosed Richter's transformation of CLL/SLL or other transformation of an indolent lymphoma, including from WM
* Subjects must not have evidence of rapidly progressive disease that would preclude subject from completing at least 1 cycle of treatment.
* Adequate organ function
* White blood cell count of ≤20 × 109/L
* Platelet count ≥30,000/uL

Exclusion Criteria:

• Disease related:

* Burkitt Lymphoma, primary central nervous system (CNS) lymphoma, Richter's transformation to Hodgkin lymphoma
* Subjects with WM who underwent plasmapheresis <35 days prior to the first dose of NKX019
* Subjects with NHL with any evidence of active CNS malignancy
* Subjects with B-ALL who have extramedullary disease (EMD)
* Subjects with any prior cellular therapy except subjects enrolling in selected cohorts who must have received prior CAR T therapy, recent HCT, or complications from HCT
* Recent use of any cancer-directed therapy within protocol specified window prior to the first dose of NKX019
* Residual toxicities ≥Grade 2 due to prior therapy
* Other comorbid conditions and concomitant medications prohibited as per study protocol
* Pregnant or lactating female

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 150 (Estimated)
Dates: Start 2021-08-20 (Actual); Primary Completion 2025-03 (Estimated); Study Completion 2038-12 (Estimated)

PRIMARY OUTCOMES:
Incidence of Treatment-Emergent Adverse Events [Safety and Tolerability] | 30 days after last dose of NKX019
  Incidence, nature, and severity of treatment related adverse events will be evaluated. An adverse event is any unfavorable and unintended sign including clinically significant abnormal laboratory findings, symptom or disease.
Proportion of subjects experiencing dose-limiting toxicities of NKX019 | 28 days from first dose of NKX019
  DLTs are defined as adverse events attributable to NKX019 treatment that occur during Cycle 1 and meet protocol-specified criteria
Objective response rate to NKX019 in Part 2 | Primary assessment: 28 days after the first dose of NKX019 followed up to 2 years after the last dose of NKX019]
  Percentage of subjects with complete and partial response. Response to treatment will be assessed based on: Lugano classification with LYRIC refinement for subjects with NHL (except CLL/SLL and WM); 2018 iwCLL guidelines for subjects with CLL/SLL; Version 1.2020 NCCN for subjects with B-ALL; consensus criteria from the 6th International Workshop on Waldenström Macroglobulinemia for subjects with WM.

SECONDARY OUTCOMES:
Assessment of NKX019 half-life | Time Frame: 28 days from first dose of NKX019
  Time required for 50% reduction from maximum amount of circulating NKX019
NKX019 duration of persistence | Followed up to 2 years after last dose of NKX019
  Testing NKX019 in peripheral blood every 3 months after dosing to determine persistence
Evaluation of host immune response against NKX019 | Followed up to 2 years after last dose of NKX019
  Serum samples will be measured for antibodies against NKX019
Objective response rate to NKX019 in Part 1 | Primary assessment: 28 days after first dose of NKX019 followed up to 2 years after last dose of NKX019
  Percentage of subjects with complete and partial response. Response to treatment will be assessed based on: Lugano classification with LYRIC refinement for subjects with NHL (except CLL/SLL and WM); 2018 iwCLL guidelines for subjects with CLL/SLL; Version 1.2020 NCCN for subjects with B-ALL; consensus criteria from the 6th International Workshop on Waldenström Macroglobulinemia for subjects with WM.

CONTACTS AND LOCATIONS:
Overall Officials: David Shook, MD, Study Director — Nkarta, Inc.
Locations (6):
- United States (2):
  - Colorado Blood Cancer Institute, Denver, Colorado
  - The Cleveland Clinic Foundation, Cleveland, Ohio
- Australia (4):
  - Institute of Haematology, Royal Prince Alfred Hospital, Camperdown, New South Wales
  - St. Vincent's Hospital, Sydney, New South Wales
  - Royal Brisbane and Woman's Hospital, Brisbane, Queensland
  - Peter MacCallum Cancer Center, Melbourne, Victoria

IPD SHARING:
Plan to Share IPD: No